CLINICAL TRIAL: NCT03081247
Title: A Randomized, Double-Blind, Parallel-Group, 12-Week, Chronic Dosing, Multi-Center Study to Assess the Efficacy and Safety of PT010 Compared to PT009 in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Brief Title: To Assess the Efficacy and Safety of PT010 Compared to PT009 in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Internal Study team decision not to proceed.
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT010017
Record Dates: First submitted 2017-03-06; First posted 2017-03-16 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BGF 320/14.4/9.6 µg MDI BID (Experimental): Budesonide, Glycopyrronium, and Formoterol Fumarate metered dose inhaler (BGF MDI)
  Interventions: Drug: BGF 320/14.4/9.6 µg MDI
- BFF 320/9.6 µg MDI BID (Experimental): Budesonide and Formoterol Fumarate metered dose inhaler (BFF MDI)
  Interventions: Drug: BFF 320/9.6 µg

INTERVENTIONS:
Drug: BGF 320/14.4/9.6 µg MDI — Budesonide, Glycopyrronium, and Formoterol Fumarate metered dose inhaler (BGF MDI)
  Other Names: PT010
  Arms: BGF 320/14.4/9.6 µg MDI BID
Drug: BFF 320/9.6 µg — Budesonide and Formoterol Fumarate metered dose inhaler (BFF MDI)
  Other Names: PT009
  Arms: BFF 320/9.6 µg MDI BID

SUMMARY:
This is a 12-week chronic-dosing study to assess the efficacy and safety of BGF MDI compared to BFF MDI in subjects with moderate to very severe COPD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, 12-week chronic-dosing study to assess the efficacy and safety of BGF MDI compared to BFF MDI in subjects with moderate to very severe COPD. The study has a total of 7 visits over a Screening Period of up to 28 days and a Treatment Period of 12 weeks followed by a telephone follow-up call 14 days after the last dose of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed Informed Consent
* Subjects with an established clinical history of COPD
* Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) ratio must be <0.70 and FEV1 must be <80% predicted normal value
* All subjects must have been on 2 or more inhaled maintenance therapies for the management of their COPD for at least 6 weeks prior to Screening
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking
* Women of Non-childbearing potential
* Women of childbearing potential and sexually active agree to prevent pregnancy by using acceptable contraceptive methods consistently

Key Exclusion Criteria:

* Significant diseases or conditions other than COPD, which in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception
* Current diagnosis of asthma
* Uncontrolled sleep apnea
* Other Serious Respiratory Disorders
* Hospitalized due to poorly controlled COPD within 6 weeks
* Poorly Controlled COPD
* Immune deficiency and/or severe neurological disorders affecting control of the upper airway
* Hypersensitivity to β2-agonists, corticosteroids, or muscarinic anticholinergics

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-16 (Estimated); Primary Completion 2018-12-07 (Estimated); Study Completion 2018-12-07 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume area under the curve from 0 to 4 hours (AUC0-4) | Week 12

SECONDARY OUTCOMES:
Change from baseline in morning pre-dose trough FEV1 | Week 12
Peak change from baseline in inspiratory capacity | Week 12
Percentage of subjects achieving a minimally clinical important difference (MCID) of 4 units or more in St. George's Respiratory Questionnaire (SGRQ) | Week 12
Time to first clinically important deterioration (CID) in COPD | 12 weeks
Change from baseline in average daily rescue Ventolin HFA use | 12 weeks
Peak change from baseline in FEV1 | Week 12
Time to onset of action | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Director — Pearl Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. The policy and additional information can be found on astrazenecaclinicaltrials.com.